CLINICAL TRIAL: NCT00412321
Title: A Phase 1 Study of Multiple Intravenous Administrations of a Chimeric Antibody Against Interleukin-6 (CNTO 328) in Subjects With B-Cell Non-Hodgkin's Lymphoma, Multiple Myeloma, or Castleman's Disease
Brief Title: A Safety and Efficacy Study of CNTO 328 in Patients With B-Cell Non-Hodgkin's Lymphoma, Multiple Myeloma, or Castleman's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR008566; C0328T03 (Other: Centocor)
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Lymphoma, Non-Hodgkin; Multiple Myeloma; Giant Lymph Node Hyperplasia
Keywords: Lymphoma, Non-Hodgkin; Multiple Myeloma; Castleman's disease; intravenous; IL-6
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Castleman Disease | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (CNTO 328) (Experimental): Patients will receive 4 administrations of 3 mg/kg CNTO 328 every 2 weeks till Day 43.
  Interventions: Drug: CNTO 328
- Cohort 2 (CNTO 328) (Experimental): Patients will receive 4 administrations of 6 mg/kg CNTO 328 every 2 weeks till Day 43.
  Interventions: Drug: CNTO 328
- Cohort 3 (CNTO 328) (Experimental): Patients will receive 3 administrations of 12 mg/kg CNTO 328 every 2 weeks till Day 43.
  Interventions: Drug: CNTO 328
- Cohort 4 (CNTO 328) (Experimental): Patients will receive 7 administrations of 6 mg/kg CNTO 328 every week till Day 43.
  Interventions: Drug: CNTO 328
- Cohort 5 (CNTO 328) (Experimental): Patients will receive 4 administrations of 12 mg/kg CNTO 328 every 2 weeks till Day 43.
  Interventions: Drug: CNTO 328
- Cohort 6 (CNTO 328) (Experimental): Patients will receive 3 administrations of 12 mg/kg CNTO 328 every 3 weeks till Day 43.
  Interventions: Drug: CNTO 328
- Cohort 7a (CNTO 328) (Experimental): Patients responding to CNTO 328 treatment will receive 9 mg/kg CNTO 328 every 3 weeks.
  Interventions: Drug: CNTO 328
- Cohort 7b (CNTO 328) (Experimental): Patients responding to CNTO 328 treatment will receive 12 mg/kg CNTO 328 every 3 weeks as extended administration.
  Interventions: Drug: CNTO 328

INTERVENTIONS:
Drug: CNTO 328 — Patients will receive administrations of CNTO 328 with dose ranging from 3 mg/kg to 12 mg/kg weekly, every 2 or 3 weeks till Day 43 in cohorts 1 to 6. After cohort 6, if the clinical response is found to be suboptimal, the patients will receive 9 mg/kg or 12 mg/kg every 3 weeks in cohorts 7a. Participants in Cohort 7a who will experience intolerable toxicity after escalating to or receiving 12 mg/kg every 3 weeks will have the option of reverting to a dose of 9 mg/kg every 3 weeks if the investigator felt it was clinically indicated. In cohort 7b participants will receive 12 mg/kg CNTO 328 every 3 weeks.

SUMMARY:
The purpose of this study is to evaluate of the study of different CNTO 328 doses and schedules and to see if CNTO 328 has any effect on Non-hodgkin's Lymphoma, Multiple Myeloma or Castleman's disease.

DETAILED DESCRIPTION:
This research study will use a type of drug called anti-IL-6 antibody, also known as CNTO 328. An antibody is a substance in the body that fights infection. CNTO 328 is an investigational drug that has been shown to slow down tumor growth or shrink tumors when tested in animals. In a previous clinical trial in patients with multiple myeloma (blood cancer), CNTO 328 appeared to be a potent inhibitor of IL-6 . One study has been completed for kidney cancer. There are studies ongoing in humans with multiple myeloma and prostate cancer to see if CNTO 328 is safe and to see what effects it has on these types of cancer. This is an open-label, nonrandomized, dose-finding phase 1 study with CNTO 328 in patients with B- cell non-Hodgkin's Lymphoma, Multiple Myeloma, or Castleman's disease. The purpose of this study is to evaluate different doses and schedules of CNTO 328 to see which dose/schedule is safe. CNTO 328 will be given through a small tube that goes directly into your vein, called an intravenous (IV) infusion. Depending on when the patient enters the study, the patient will be assigned to receive one course of CNTO 328 in one of the following groups: Group 1: 3 mg/kg 2 hr IV infusion every 2 weeks for 4 doses. Group 2: 6 mg/kg 2 hr IV infusion every 2 weeks for 4 doses. Group 3: 12 mg/kg 2 hr IV infusion every 3 weeks for 3 doses. Group 4: 6 mg/kg 2 hr IV infusion every week for 7 doses. Group 5: 12 mg/kg 2 hr IV infusion every 2 weeks for 4 doses. Group 6: 12 mg/kg 1 hr IV infusion every 3 weeks for 3 doses. Group 7a: 9 mg/kg 1 hr IV infusion every 3 weeks. Group 7b: 12 mg/kg 1hr IV infusion every 3 weeks for Castleman's patients only. In Groups 1-5, the overall amount of study drug that will be given increases with each higher group. Group 1 will be filled before Group 2 starts and Group 2 will be filled before Group 3 starts, etc. In this way, CNTO 328 can be tested more safely. Both the patient and the study doctor will know to which group the patient is assigned. Patients will remain in the group that they are assigned to for the entire time of participation in the study. Up to 70 patients may take part in this study. Patients in Groups 1-6 will be in the study for up to 34 weeks prior to Post Study Follow-Up. Screening: up to 4 weeks before the first dose schedule of CNTO 328. Treatment: up to 6 weeks of treatment with CNTO 328. Extended Dosing: Patients assigned to Groups 1-6, and their cancer or disease has become stable or better while receiving CNTO 328, may be able to receive additional courses of study drug. Patients in Group 7 will be in the study until their disease gets worse, they can no longer tolerate CNTO 328, the study doctor feels it is in their best interest to stop CNTO 328 or they longer wish to participate in the study. Long Term Follow-Up: Patients will be contacted by telephone every six months after the last infusion of study drug to assess the patient's disease status and survival. Dose (6-12 mg/kg) and frequency (weekly or 2 or 3 week intervals) of dosing depends upon Group assignment. CNTO 328 will be given through a small tube that goes directly into your vein, called an intravenous (IV) infusion. The infusion will take about 2 hours to complete for groups 1-5 and 1 hour for Groups 6 and 7. In Groups 1-6, CNTO 328 will be given once every 1, 2 or 3 weeks from days 1 to 43 depending on treatment assignment. In Group 7a and Group 7b, CNTO 328 will be given on day 1 of each 21 day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with B-cell non-Hodgkin's lymphoma, multiple myeloma, or Castleman's Disease which has progressed on or after standard therapy or for which there is no effective standard therapy, or which is not suitable for standard therapy
* Detectable serum C-Reactive Protein
* At least 4 weeks since prior systemic therapy, radiotherapy, or surgery
* Must meet protocol lab criteria (adequate bone marrow, liver and renal function) to be assessed at patient's first visit to the study center

Exclusion Criteria:

* Received any investigational drug within 30 days or 5 half-lives of the investigational drug, whichever is longer
* History of receiving murine or human-murine recombination products, such as G250, BE-8, and other monoclonal antibodies. (Note: Prior rituximab treatment is not an exclusion criterion)
* Serious concurrent illness or significant cardiac disease characterized by significant ischemic coronary disease or congestive heart failure
* Known human immunodeficiency virus seropositivity, acquired immunodeficiency syndome, hepatitis C or active hepatitis B infection. For Cohort 7, known human herpesvirus-8 seropositivity
* Presence of a transplanted solid organ (with the exception of a corneal transplant more than 3 months prior to screening) or having received an allogeneic bone marrow transplant or an allogeneic peripheral blood stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Adverse Events as a Measure of Safety and Tolerability | Up to 3 years after the last administration of study medication
  Number of Patients with adverse events will be reported.
Serum Concentration of CNTO 328 | Up to Day 71
  Serum Concentration of CNTO 328 will be reported.

SECONDARY OUTCOMES:
Pharmacodynamics of CNTO 328 | Up to Day 71
  Pharmacodynamic parameters C-reactive protein, interleukin-6 (IL-6), soluble IL-6 receptor [GP80], soluble GP130, TNFα, ΙL-8, IL-10, soluble IL-2 receptor (sIL-2R), IFNγ, serum amyloid A (SAA), N-telopeptide (NTx), C-telopeptide (CTx), hepcidin-25, VEGF, and fibroblast growth factor will be assessed.
Plasma antibodies to CNTO 328 | Up to Week 24
  Plasma antibodies to CNTO 328 will be used to evaluate the immunogenicity of CNTO 328.
Number of participants with Castleman's disease who achieved tumor response | Screening phase (4 weeks before administration of study medication), Day 36, and Day 57
  Evaluation of tumor response for subjects with Castleman's disease were performed by central review according to the standard criteria, developed by an NCI-sponsored international working group (Cheson et al, 1999).
Number of participants with multiple myeloma who achieved disease response | Screening phase (4 weeks before administration of study medication), Day 36, and Day 57
  Evaluation of disease response for subjects with Multiple Myeloma were performed by the investigators according to the response criteria developed by an international group of multiple myeloma and bone marrow transplant experts (Blade et al, 1998).
Number of participants with B-cell non-Hodgkin's lymphoma and multiple myeloma who achieved clinical benefit (CB) | Up to Day 71
  CB will assess pain (by Pain intensity [PI] and 7-items assessing how much pain interfered with daily activities), performance status (by Karnofsky performance status which quantifies participant's well-being and activities of daily life), and weight change. PI score will be assessed by 4 questions (Q) rated on 11-point numerical rating scale ranging from "0=no pain" to "10=higher severity of pain". Each participant will be classified as either CB responder (i.e., if +ve for at least 1 of 3 primary CB measures and stable for other 2) or Non-responder (If a participant is stable on all 3 primary measures OR if -ve for any 1 of 3 primary measures).
Number of participants with Castleman's disease who achieved clinical benefit | Up to Day 71
  CB assessments for participant with Castleman's disease consist of the following 6 measures: hemoglobin, fatigue, anorexia, fever, weight, and size of largest lymph node. Each participant will be classified as either improved, stable, or worsening for each of the measures. If a participant has improved for at least 1 of the 6 measures and is at least stable for the remaining measures, participant will be considered to be a responder for CB. If a participant has worsening for at least 1 of the 6 measures, participant will be considered as having progression for CB. Any other participant will be considered to be stable for CB. Any "improved" or "stable" assessment of the lymph node parameter for CB must be confirmed by radiographic imaging. If a participant shows progression for CB at 2 consecutive assessments the participant must discontinue study treatment.
Number of participants with B-cell non-Hodgkin's lymphoma who achieved disease response | Screening phase (4 weeks before administration of study medication), Day 36, and Day 57
  Evaluation of disease response for subjects with B-cell non-Hodgkin's lymphoma were performed by the investigators according to the standard criteria, developed by an NCI-sponsored international working group (Cheson et al, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (9):
- United States (9):
  - Little Rock, Arkansas
  - Tampa, Florida
  - Atlanta, Georgia
  - Box 302, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington

REFERENCES:
- See also: A Phase 1 Study of Multiple Intravenous Administrations of a Chimeric Antibody Against Interleukin-6 (CNTO 328) in Subjects with B-Cell Non-Hodgkin's Lymphoma, Multiple Myeloma, or Castleman's Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=171&filename=CR008566_CSR.pdf